CLINICAL TRIAL: NCT05247307
Title: Clinical Efficacy of the Infusion of Donor Plasma, Convalescent From SARS-CoV-2 Infection, to Patients With Recent Infection.
Brief Title: Efficacy of the Infusion of Donor Plasma in COVID-19 Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy of treatment tested
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Jose Enrique de la Puerta, MD, Principal Investigator, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SARS VOC 2 GALDAKAO 02
Record Dates: First submitted 2022-02-17; First posted 2022-02-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: COVID-19; Clinical Trial Protocol; Immunization, Passive
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1; experimental group: control group), double-blind study, in which the doctors who prescribe the treatments and those who assess the results do not know the treatment received by the patient.
  The convalescent plasma will be contrasted with fresh frozen plasma, available at the Basque Transfusion and Tissue Center of the Basque Autonomous Community (CVTTH), obtained before 12/31/2019.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment in the intervention group:
  Infusion of 300 cc of convalescent donor plasma from COVID 19, administered within more than 168 hours from the onset of symptoms
  Treatment in the control group:
  For the study to be blind, the infusion of non-convalescent donor plasma, obtained before the start of the epidemic, is required to guarantee the absence of anti-COVID antibodies in the plasma of the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Treatment in the intervention group:
  Infusion of 300 cc of convalescent donor plasma from COVID 19, administered within more than 168 hours from the onset of symptoms Treatments in both arms of the study All patients included in the study will receive the same standard treatment that is deemed appropriate at any time, understanding as standard treatment that established at any time by the guidelines established by the Department of Health, or by the Osakidetza Directorate, in each moment.
  Interventions: Biological: convalescent plasma infusion covid 19
- Control (Active Comparator): Treatment in the control group:
  For the study to be blind, the infusion of non-convalescent donor plasma, obtained before the start of the epidemic, is required to guarantee the absence of anti-COVID antibodies in the plasma of the control group.
  Treatments in both arms of the study All patients included in the study will receive the same standard treatment that is deemed appropriate at any time, understanding as standard treatment that established at any time by the guidelines established by the Department of Health, or by the Osakidetza Directorate, in each moment.
  Interventions: Biological: convalescent plasma infusion covid 19

INTERVENTIONS:
Biological: convalescent plasma infusion covid 19 — Operating process
  * A single dose of plasma (300 mL) immune anti-coronavirus or not, depending on what corresponds will be infused.
  * The collaborating staff will enter the initial and follow-up data in Red Cap based on the information contained in the medical record, or by talking to the patient by telephone to clarify any doubts.

SUMMARY:
Objectives Primary objectives To assess the superiority or not of the infusion of anti-COVID immune plasma infusion versus a placebo (non-immune plasma) to patients over 65 years of age recently infected with the SARS-CoV-2 coronavirus, to prevent progression to severe forms of the disease with hospital admission.

Secondary objectives To assess if the intervention improves the clinical evolution of the target patient.

* Improvement of the disease.
* Disease deterioration Methodology Design Prospective, randomized (1:1; experimental group: control group), double-blind study, in which the doctors who prescribe the treatments and those who assess the results do not know the treatment received by the patient.

Methods. Patients 65 years of age or older will be included, diagnosed with SARS-CoV-2 coronavirus infection, in which no more than 7 days have elapsed since the onset of symptoms or diagnosis to plasma infusion.All patients included in the study will receive the same standard treatment that is deemed appropriate at any time, understanding as standard treatment that established at any time by the guidelines established.Infusion of 300 cc of convalescent donor plasma from COVID 19, administered within more than 168 hours from the onset of symptoms. For the study to be blind, the infusion of non-convalescent donor plasma, obtained before the start of the epidemic, is required to guarantee the absence of anti-COVID antibodies in the plasma of the control group.

Analysis of data:

Initially, the homogenization of the data referring to the two groups of studies will be evaluated. Classical statistical tests will be applied, such as Wilcoxon's non-parametric tests for the comparison of means of continuous variables, as well as the Chi-square test (or Fisher's exact test) to evaluate the association between categorical variables. The result variables are:

1. Hospital admission
2. Clinical course
3. Mortality
4. Complications and/or adverse effects of plasma.

DETAILED DESCRIPTION:
Objectives Primary objectives To assess the superiority or not of the infusion of anti-COVID immune plasma infusion versus a placebo (non-immune plasma) to patients over 65 years of age recently infected with the SARS CoV 2 coronavirus, to prevent progression to severe forms of the disease with hospital admission.

Secondary objectives To assess if the intervention improves the clinical evolution of the target patient.

* Improvement of the disease is considered decrease in the WHO scale.
* Disease deterioration is considered ascent of the WHO scale
* It is considered stable disease those cases in which criteria for improvement or deterioration of the disease are not met.

Methodology Design Prospective, randomized (1:1; experimental group: control group), double-blind study, in which the doctors who prescribe the treatments and those who assess the results do not know the treatment received by the patient.

The convalescent plasma will be contrasted with fresh frozen plasma, available at the Basque Transfusion and Tissue Center of the Basque Autonomous Community (CVTTH), obtained before 12/31/2019.

Sample size for the main objective To calculate the sample size, it is assumed that the hospital admission rate in this age group is 17%, obtained from the Galdakao Hospital database during the second peak of the pandemic (from 6/15/2020 to 9/8/2020).

The following variables are assumed:

* There is only one experimental arm
* Ratio cases: controls: 1:1
* Proportion in reference group: >17%
* Proportion in the intervention group: ≤ 5%
* Type I Error (alpha): 5%
* Power: 80%
* Loss ratio: 10%
* N reference group: 100
* N intervention group: 100 Accepting an alpha risk of 0.05 and a power of 0.8 in a bilateral contrast, 91 subjects are needed in the first group and 91 in the second to detect as statistically significant the difference between two proportions, which for group 1 is expected to be the proportion of admitted patients is more than 17 in the control group and 5% or less in the intervention group, for which, assuming a percentage of losses of no more than 10% in follow-up, at least 100 patients in each branch. The arcsine approximation has been used.

Data analysis and interim study For the calculation of the results, the Statistical Analysis System (SAS) application will be used, calculating the difference in the proportion for the objectives, the relative risk, as well as its statistical significance.

A first interim analysis will be carried out after the entry of 50% of the cases necessary for hospital admission (93 cases without previous admission). In the event that a statistically significant difference (p=0.05) has been achieved for the immune plasma arm, the modification of the distribution ratio of patients between both arms (adaptive study) will be assessed, or the interruption of the study if so. deems appropriate. In the event that significant unexpected adverse effects are observed, the study will be discontinued.

Likewise, at the end of the study, an analysis of the variables related to the result (prognostic data at diagnosis) will be carried out, using multiple linear regression analysis.

Study patients and plasma donors Patients 65 years of age or older will be included, diagnosed with SARS-CoV-2 coronavirus infection, in which no more than 7 days have elapsed since the onset of symptoms or diagnosis to plasma infusion.

Inclusion criteria:

* SARS-CoV-2 infection, confirmed by polymerase chain reaction amplification (PCR) or technique of similar specificity.
* Symptom onset, or positive PCR (whichever comes first) within 7 days (168 hours) prior to planned plasma infusion.
* 65 years of age or older.
* All patients, or the guardian appointed by the judge, in the case of recognized judicial incapacity, must sign the informed consent document.

Exclusion criteria:

* Less than 65 years of age
* Symptom onset, or positive PCR (whichever comes first), more than 7 days (168 hours) prior to planned plasma infusion.
* Severe dementia, or other significant comorbidity, that generates a serious deterioration of the baseline functional status, with a life expectancy of less than 6 months.
* Participation in another clinical trial or study.
* History of allergy to amotosalen or psoralens Donor selection and plasmapheresis

For the selection of donors and plasmapheresis, the recent criteria developed by the Scientific Committee for Transfusion Safety (CCST) of the Ministry of Health Version 2.0 - April 15, 2020 "RECOMMENDATIONS FOR OBTAINING PLASMA FROM CONVALESCENT COVID-19 DONORS" are adopted. Donors will meet the standard criteria for blood donation, except the recent diagnosis of SARS-CoV-2 infection, and in addition the following:

1. Signed the specific informed consent document for donation for the trial. In the event that the trial becomes multicenter, the plasma of the donors recruited by each center will be reserved for the patients included in it, unless expressly agreed by the centers involved for specific cases.
2. Having had a SARS-CoV-2 infection in the last 3 months, confirmed by PCR or a technique of similar specificity.
3. Those cases that have presented a mild infection, without confirmation by PCR, but that meet criterion 7 may be included.
4. Meet both criteria:

   1. Minimum of 14 days without symptoms
   2. At least one negative PCR for viral RNA in the upper respiratory tract.
5. Not having received corticosteroids in the last week.
6. Presence of anti-COVID-19 immunoglobulin G ( IgG) antibodies by immunoassay or similar reliability.
7. Those who have reached 18 years of age and preferably under 60 years of age, although in the event of de-provisioning it is considered that the age range can be extended to 65 years of age, provided that the general condition of the donor allows it.
8. Preferably they will be men who have never been transfused.
9. The plasma obtained from the donor will be, whenever possible, subjected to inactivation treatment or quarantine.
10. The donor will sign the standard informed consent document for the donation of plasma from the Basque Center for Transfusion and Human Tissues of the Basque Autonomous Community.

The INTERCEPT™ Blood System for Plasma is used for plasma inactivation. The system uses a solution of amotosalen.

Intervention Treatments in both arms of the study All patients included in the study will receive the same standard treatment that is deemed appropriate at any time, understanding as standard treatment that established at any time by the guidelines established by the Department of Health, or by the Osakidetza Directorate, in each moment.

Treatment in the intervention group:

Infusion of 300 cc of convalescent donor plasma from COVID 19, administered within more than 168 hours from the onset of symptoms

Treatment in the control group:

For the study to be blind, the infusion of non-convalescent donor plasma, obtained before the start of the epidemic, is required to guarantee the absence of anti-COVID antibodies in the plasma of the control group.

Monitoring, recording and communication of Adverse Events (AA), Adverse Drug Reactions (ADR), and Serious Adverse Event (SAE) Any detrimental medical event that occurs in a patient to whom the plasma has been administered, although not necessarily causally related to such treatment, will be monitored, recorded, and reported. The physician must record in the medical record all AEs, ADRs, and SAEs that occur from the time the patient signed the informed consent until 28 days have elapsed after the patient's last follow-up visit within the study. Evaluation of adverse events: a qualified physician will assess all adverse events with respect to their severity. The adverse effects observed will be communicated by the usual haemovigilance means established by Law (ROYAL DECREE 1088/2005, of September 16, which establishes the technical requirements and minimum conditions for blood donation and transfusion centers and services). Additionally, the adverse effects observed will be reported to the Spanish Agency for Medicines and Health Products.

Operating process

* A single dose of plasma (300 mL) immune anti-coronavirus or not, depending on what corresponds will be infused.
* The collaborating staff will enter the initial and follow-up data in Red Cap based on the information contained in Osabide, or by talking to the patient by telephone to clarify any doubts.

Prognostic variables to collect for each case

Baseline data at study entry (prior to plasma infusion):

* Age at diagnosis of SARS CoV 2 infection
* Sex
* Associated diseases:

  * Hypertension
  * Diabetes
  * Cerebrovascular disease
  * chronic obstructive pulmonary disease (COPD)
* Hospital admission prior to plasma infusion due to complications of infection (COVID--19) (Y/N)
* Analytical prognostic factors:
* Neutrophils
* Lymphocytes
* D-dimers
* Urea
* lactate dehydrogenase (LDH)
* glutamate oxaloacetate transaminase (GOT)
* glutamate-pyruvate transaminase (GPT)
* Total bilirubin
* Troponin T
* Procalcitonin
* PCR
* Ferritin
* Case code
* WHO Scale Plasma infusion data
* Date of infusion
* Infusional reaction (Y/N)
* Data of the infusional reaction (if applicable)
* Period of donor infection in case of immune plasma
* Plasma type (immune; control)
* Neutralizing antibody titer Evolutionary variables to collect for each case On days +7, +14, +28, and +120 post plasma infusion (28 days for hospital admission or clinical evolution, and 120 days for mortality)

  * Date (of recorded data)
  * Clinical situation (WHO scale) on the 7th, 14th, and 28th day after plasma infusion
  * Admitted to hospital (Y/N) Analytical profile days +7, +14, and +28 following the infusion.
* Neutrophils
* Lymphocytes
* D-dimers
* Urea
* lactate dehydrogenase (LDH)
* glutamate oxaloacetate transaminase (GOT)
* glutamate-pyruvate transaminase (GPT)
* Total bilirubin
* Troponin T
* Procalcitonin
* PCR
* Ferritin Final data (day +28; day +120 for mortality)
* data date
* Specific anti-COVID 19 treatment received, in addition to plasma.
* Deceased (Y/N)
* Date of death in your case
* Entered (Y/N)
* Date of entry in your case
* Date of discharge in your case
* Reason for discharge (healed or improved; deceased; other) ANALYSIS OF DATA Initially, the homogenization of the data referring to the two groups of studies will be evaluated. Classical statistical tests will be applied, such as Wilcoxon's non-parametric tests for the comparison of means of continuous variables, as well as the Chi-square test (or Fisher's exact test) to evaluate the association between categorical variables.

The result variables are:

1. Hospital admission (among patients whose admission was not indicated prior to plasma infusion
2. Clinical course: Improvement / stable / deterioration of the disease on the 7th and 14th days after plasma infusion.
3. Mortality (in-hospital and out-of-hospital)
4. Complications and/or adverse effects of plasma. To determine the predictive factors of hospital admission, Poisson regression and/or negative binomial models will be developed, following the same procedure mentioned above.

All calculations will be performed with the SAS System v9.4 statistical package and statistical significance will be considered when p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* SARS CoV 2 infection, confirmed by PCR or technique of similar specificity.
* Symptom onset, or positive PCR (whichever comes first) within 7 days (168 hours) prior to planned plasma infusion.
* 65 years of age or older.
* All patients, or the guardian appointed by the judge, in the case of recognized judicial incapacity, must sign the informed consent document.

Exclusion Criteria:

* Less than 65 years of age
* Symptom onset, or positive PCR (whichever comes first), more than 7 days (168 hours) prior to planned plasma infusion.
* Severe dementia, or other significant comorbidity, that generates a serious deterioration of the baseline functional status, with a life expectancy of less than 6 months.
* Participation in another clinical trial or study.
* History of allergy to amotosalen or psoralens

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of hospital admission | 28 days
  Rate of hospital admission (among patients whose admission was not indicated prior to plasma infusion
Rate of severity of the disease | 28 days
  Rate of improvement / stable / deterioration of the disease on the 7th and 14th days after plasma infusion.
Rate of of deaths | 120 days
  Rate of of deaths (in-hospital and out-of-hospital)
Rate of complications | 28 days
  Rate of complications and/or adverse effects of plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Enrique de la Puerta Rueda, MD, Principal Investigator — Hospital Cruz Roja de Bilbao; Maria Cristina Martinez Bilbao, MD, Principal Investigator — Hospital Universitario Galdakao Usansolo; Amaia Uresandi Iruin, MD, Principal Investigator — Hospital Universitario de Cruces
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Around this year 2022
Access Criteria: Contact with principal investigator